CLINICAL TRIAL: NCT02480023
Title: Changes in Bone Mineral Density as Measured by Calcaneal Quantitative Ultrasound in Third Trimester of Pregnancy
Brief Title: Assessment of Bone Mineral Density During Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, Prof. Mohamed Laban, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: osteopenia during pregnancy
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Bone Mineral Density Quantitative Trait Locus 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- healthcare (Experimental): QUS for calcaneus bone of right foot will be done for this group of Pregnant women at the third trimester
  Interventions: Radiation: calcaneal quantitative ultrasound assessment

INTERVENTIONS:
Radiation: calcaneal quantitative ultrasound assessment — QUS for calcaneus bone of right foot will be done for this group of Pregnant women at the third trimester

SUMMARY:
BMD at peripheral sites typically heel is measured by Ultrasound densitometry at Ain Shams Maternity hospital.

DETAILED DESCRIPTION:
Consecutive patients with singleton pregnancies between 36 and 39 weeks booked at a general obstetric clinic in a regional hospital will be recruited for the study. The obstetric department is a tertiary referral center in the region and part of a university teaching unit which catered to an annual delivery of around 10,000 women. A group of first trimester pregnant women with nearly the same age is recruited as controls.

ELIGIBILITY:
Inclusion Criteria:

1. females during 3rd trimister

Exclusion Criteria:

1. Secondary causes of bone loss such as hyperparathyroidism.
2. Co-morbidities that would interfere with bone metabolism as clinically significant liver or renal disease.
3. Physical or orthopedic disabilities that would place the subject at risk or limit their ability to perform US.
4. Taking medication known to affect bone including steroid hormones.

Histories of smoking and use of oral contraceptives (OCs) are not exclusion criteria.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density loss during pregnancy that is detectable by quantitative ultrasound at the os calcis. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: mohamed laban, MD, Study Chair — Ain Shams University
Locations (1):
- Faculty of medicine, ain shams university, Cairo, Cairo Governorate, Egypt